CLINICAL TRIAL: NCT02215161
Title: Phase II Single Agent Study of Selinexor (KPT-330) in Patients With Metastatic Castration-Resistant Prostate Cancer (mCRPC) and Prior Therapy With Abiraterone and/or Enzalutamide
Brief Title: Selinexor in Treating Patients With Abiraterone Acetate and/or Enzalutamide Refractory Metastatic Castration-Resistant Prostate Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Risk to benefit ratio is not acceptable
Sponsor: University of California, San Francisco (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14552; NCI-2014-01936 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 14-13390; 14552 (Other: University of California, San Francisco)
Record Dates: First submitted 2014-07-30; First posted 2014-08-13 (Estimated); Results first posted 2018-06-26 (Actual); Last update posted 2018-06-26 (Actual); Status verified 2018-05

CONDITIONS: Castration Levels of Testosterone; Hormone-Resistant Prostate Cancer; Metastatic Prostate Carcinoma in the Soft Tissue; Prostate Carcinoma Metastatic in the Bone; PSA Progression; Stage IV Prostate Adenocarcinoma AJCC v7
MeSH Terms: interventions — selinexor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (selinexor) (Experimental): Patients receive selinexor PO on days 1 and 3 of weeks 1-3. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Selinexor

INTERVENTIONS:
Drug: Selinexor — Given PO
  Other Names: CRM1 Nuclear Export Inhibitor KPT-330; KPT-330; Selective Inhibitor of Nuclear Export KPT-330; SINE KPT-330

SUMMARY:
This phase II trial studies selinexor in treating patients with prostate cancer that has spread to other parts of the body (metastatic), keeps growing even when the amount of testosterone in the body is reduced to very low levels (castration-resistant), and did not respond to treatment (refractory) with abiraterone acetate and/or enzalutamide. Selinexor may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To describe radiographic progression free survival (rPFS) associated with selinexor in patients with abiraterone (abiraterone acetate) refractory metastatic castration-resistant prostate cancer (mCRPC).

SECONDARY OBJECTIVES:

I. To measure prostate-specific antigen (PSA) changes at 12 weeks post-selinexor initiation.

II. To assess time to PSA progression. III. To measure time to development of >= 2 new bone lesions. IV. To compare the relationship of abiraterone-resistance status (primary vs acquired) and treatment outcome.

V. To determine the effect of selinexor on persistent pain associated with bone metastasis using the brief pain inventory (BPI) short form.

VI. To describe the safety profile of selinexor in patients with metastatic castration-resistant prostate cancer.

VII. To determine the effect of selinexor on circulating leukocyte exportin 1 (XPO-1) expression, leukocyte gene expression profile and macrophage inhibitory cytokine-1 (MIC-1) messenger ribonucleic acid (mRNA) expression.

VIII. To assess serum selinexor trough levels as a function of dose and time since last dose.

TERTIARY OBJECTIVES:

I. To describe the relationship of XPO-1 expression to PSA decline. II. To describe the expression profile of metastatic tumor and outcome. III. To describe the type of progression (e.g. pain, bone etc). IV. To define XPO-1 expression in patients for whom pre- and post-treatment biopsy is obtained.

OUTLINE:

Patients receive selinexor orally (PO) on days 1 and 3 of weeks 1-3. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 30 days and then every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the prostate
* Patients must have castrate levels of testosterone (< 50 ng/dL) on gonadotropin-releasing hormone (GnRH) analogues or have had prior orchiectomy; GnRH analogues must be continued while on study
* Tumor tissue submitted for molecular and genetic analysis through the companion Stand-up 2 Cancer (SU2C) radiologically guided biopsy of abiraterone and/or enzalutamide refractory mCRPC protocol

  * Patients who consent to participate in the companion biopsy protocol and are subsequently determined to be ineligible for biopsy are eligible to participate in the current protocol
* Progressive disease as demonstrated by a rising PSA (at least two determinations) prior to study entry, and/or radiographic evidence of tumor progression in soft tissue according to modified Response Evaluation Criteria In Solid Tumors (RECIST) criteria or identification of new lesions by bone scan (i.e., >= 2 new lesions)
* Primary resistance or acquired resistance (i.e., acquired resistance will be defined as disease progression following a period of response defined as >= 50% decline in PSA within 12 weeks of starting therapy and not otherwise meeting criteria for primary resistance) to any of the following agents/combinations of therapy:
* Abiraterone acetate; primary resistance to abiraterone will be defined as:

  * No PSA decline
  * PSA decline less than 50% after 12 weeks of abiraterone therapy
  * PSA progression within 12 weeks of abiraterone acetate (AA) treatment (by Prostate Cancer Working Group-2 [PCWG2] criteria), after initial response to therapy
  * Objective progression, by RECIST criteria for soft tissue lesions and by modified PCWG2 criteria for bone lesions within 12 weeks of starting abiraterone treatment
  * Unequivocal clinical progression (per the treating provider's discretion) within 12 weeks of starting abiraterone treatment
* Enzalutamide; primary resistance to enzalutamide will be defined as:

  * No PSA decline
  * PSA decline less than 50% after 12 weeks of enzalutamide therapy
  * PSA progression within 12 weeks of enzalutamide treatment (by PCWG2 criteria), after initial response to therapy
  * Objective progression, by RECIST criteria for soft tissue lesions and by modified PCWG2 criteria for bone lesions within 12 weeks of starting enzalutamide treatment
  * Unequivocal clinical progression (per the treating provider's discretion) within 12 weeks of starting enzalutamide treatment
* Other second-generation investigational anti-androgen/androgen-receptor targeted therapies, including apalutamide (ARN-509); primary resistance will be defined as:

  * No PSA decline
  * PSA decline less than 50% after 12 weeks of enzalutamide therapy
  * PSA progression within 12 weeks of enzalutamide treatment (by PCWG2 criteria), after initial response to therapy
  * Objective progression, by RECIST criteria for soft tissue lesions and by modified PCWG2 criteria for bone lesions within 12 weeks of starting enzalutamide treatment
  * Unequivocal clinical progression (per the treating provider's discretion) within 12 weeks of starting enzalutamide treatment
* Combination therapy with abiraterone, enzalutamide and/or other second- generation investigational anti-androgen/androgen-receptor targeted therapies, including ARN-509; primary resistance to combination therapy will be defined as:

  * No PSA decline
  * PSA decline less than 50% after 12 weeks of abiraterone and enzalutamide therapy
  * PSA progression within 12 weeks of abiraterone and enzalutamide treatment (by PCWG2 criteria), after initial response to therapy
  * Objective progression, by RECIST criteria for soft tissue lesions and by modified PCWG2 criteria for bone lesions within 12 weeks of starting abiraterone and enzalutamide treatment
  * Unequivocal clinical progression (per the treating provider?s discretion) within 12 weeks of starting abiraterone and enzalutamide treatment
* Sequenced therapy, including any of the following:

  * Abiraterone acetate followed by enzalutamide

    * Primary resistance will be defined per criteria for abiraterone monotherapy primary resistance
  * Enzalutamide followed by abiraterone acetate

    * Primary resistance will be defined per criteria for enzalutamide monotherapy primary resistance
  * Other second-generation investigational anti-androgen/androgen- receptor targeted therapies, including ARN-509

    * Primary resistance will be defined per criteria for other investigational anti-androgen monotherapy primary resistance
* Presence of 1 or more bone metastasis
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Prior and ongoing zoledronic acid or denosumab therapy is allowed
* Prior therapy with radium-223 is allowed
* Discontinuation of prior therapy for mCRPC: a washout period of 28 days for the following therapies is required: abiraterone, enzalutamide, fluconazole, itraconazole, flutamide, bicalutamide, nilutamide, and other experimental hormonal agents (ARN509, orteronel [TAK-700], etc.), sipuleucel-T (Provenge), other experimental vaccines (PROSTVAC-V/F, etc.), strontium-89, samarium, and radium-223 chloride
* Leukocytes > 3,000/mcL
* Absolute neutrophil count > 1,500/mcL
* Platelets > 125,000/mcL
* Hemoglobin >= 5.59 mmol/L or 9 g/dL; up to 5% deviation is tolerated; transfusions and growth factors are allowed
* Total bilirubin within normal institutional limits
* Aspartate aminotransferase (AST)(serum glutamic oxaloacetic transaminase [SGOT]) < 3 X institutional upper limit of normal
* Alanine aminotransferase (ALT)(serum glutamate pyruvate transaminase [SGPT]) < 3 X institutional upper limit of normal
* Creatinine within normal institutional limits OR creatinine clearance > 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Ability to understand a written informed consent document, and the willingness to sign it
* Life expectancy of at least 12 weeks
* Able to swallow and retain oral medication

Exclusion Criteria:

* Untreated brain metastases; brain metastases =< 1 cm and not associated with any focal neurologic deficits are allowed
* Prior docetaxel or other chemotherapy for mCRPC; patients who have received docetaxel for metastatic hormone-sensitive prostate cancer are eligible
* Active or symptomatic viral hepatitis or chronic liver disease
* Clinically significant heart disease as evidenced by myocardial infarction, or arterial thrombotic events in the past 6 months, severe or unstable angina, or New York Heart Association (NYHA) class II-IV heart disease or known cardiac ejection fraction measurement of < 50 % at baseline
* Patients with significantly diseased or obstructed gastrointestinal tract or uncontrolled vomiting or diarrhea or other gastrointestinal disorders (medical disorders or extensive surgery) that may interfere with the absorption of the study agents
* Pure small cell carcinoma of the prostate or any mixed histology cancer of the prostate (eg: neuroendocrine) that contains < 50% adenocarcinoma, as observed on biopsy obtained at the time of diagnosis or on any subsequent biopsies
* Any ?currently active? second malignancy, other than non-melanoma skin cancer; patients are not considered to have a "currently active? malignancy, if they have completed therapy and are considered by their physician to be at least less than 30% risk of relapse over next year
* Any condition, which in the opinion of the investigator, would preclude participation in this trial
* Active psychiatric illnesses/social situations that would limit compliance with protocol requirements
* Patients in whom urgent treatment with docetaxel is indicated, per clinician discretion; this includes, but is not limited to patients with symptomatic visceral metastatic disease
* Uncontrolled infection or concomitant medical illness that is not adequately controlled with current medical management, as determined per clinician discretion
* Active bleeding disorders or evidence of evidence of chronic or acute disseminated intravascular coagulation (DIC)
* Severely compromised immunological state, including known human immunodeficiency virus (HIV)
* Any acute toxicities due to prior anti-cancer treatments and/or radiotherapy that have not resolved to a National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) grade of =< 1 (except alopecia)
* Prior radiation therapy completed < 3 weeks or single fraction of palliative radiotherapy < 14 days prior to first dose of KPT-330 (selinexor)
* Initiation of bisphosphonate therapy < 4 weeks prior to first dose of KPT-330; patients receiving bisphosphonate or denosumab therapy must be on stable doses for at least 4 weeks prior to first dose of KPT-330
* Men unable or unwilling to employ 2 forms of highly effective contraception throughout the study and for 8 weeks after the end of study treatment

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2014-09-02 (Actual); Primary Completion 2017-02-15 (Actual); Study Completion 2018-04-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Ryan, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

REFERENCES:
- [Derived] Wei XX, Siegel AP, Aggarwal R, Lin AM, Friedlander TW, Fong L, Kim W, Louttit M, Chang E, Zhang L, Ryan CJ. A Phase II Trial of Selinexor, an Oral Selective Inhibitor of Nuclear Export Compound, in Abiraterone- and/or Enzalutamide-Refractory Metastatic Castration-Resistant Prostate Cancer. Oncologist. 2018 Jun;23(6):656-e64. doi: 10.1634/theoncologist.2017-0624. Epub 2018 Feb 27. PMID 29487219

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Selinexor): BID: twice a day D: day PO: oral 1 cycle = 4 weeks, 28 days
  Premedication:
  * Ondansetron 8 mg PO every 8 hours on day prior to and day of dosing (D0-D3)
  * Olanzapine 5 mg PO at bedtime or 2.5 mg PO BID on day of dosing (D1, D3)
  Study drug:
  - Selinexor PO on D1 and D3 of weeks 1-3 of each cycle. Drug holiday on week 4. Courses repeat every 28 days in absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Treatment (Selinexor)
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Selinexor)
Number analyzed (Participants) | 14
Age, Customized [Count of Participants; unit: Participants]
  Age Group: 50 - 59 | 1
  Age Group: 60 - 69 | 3
  Age Group: 70 - 79 | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 11
  More than one race | 1
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Radiographic Progression Free Survival (rPFS)
Description: Defined as the time from study start until one of the following events occurs: >= 2 new bone lesions on technetium bone scan; Response Evaluation Criteria in Solid Tumors (RECIST)-defined tumor progression; clinical deterioration requiring a change in prostate cancer therapy, or at clinician discretion; surgery or radiation to treat a prostate cancer related indication; or death from any cause.
Time Frame: From study start up to 3 years
Measure: Median (Full Range); unit: weeks
Groups:
- Treatment (Selinexor): BID: twice a day D: day PO: oral 1 cycle = 4 weeks, 28 days
  Premedication:
  * 8mg Ondansetron PO every 8 hours on day prior to and day of dosing (D0-D3)
  * 5mg Olanzapine PO at bedtime or 2.5 mg PO BID on day of dosing (D1, D3)
  Study drug:
  - 60mg Selinexor PO on D1 and D3 of weeks 1-3 of each cycle. Drug holiday on week 4. Courses repeat every 28 days in absence of disease progression or unacceptable toxicity.
Arm/Group | Treatment (Selinexor)
Number analyzed (Participants) | 14
weeks | 31 [7 to 47]

2. Secondary Outcome: Abiraterone Resistance Status (Primary Versus Acquired)
Description: Comparison of radiographic progression free survival between patients with primary abiraterone resistance and acquired abiraterone resistance using a Cox proportional hazards model.
Time Frame: At baseline
Population: The study was terminated due to unacceptable toxicity. Data on resistance type was not collected.
Groups:
- Primary Abiraterone Resistance; Aquired Abiraterone Resistance: BID: twice a day D: day PO: oral 1 cycle = 4 weeks, 28 days
  Premedication:
  * 8mg Ondansetron PO every 8 hours on day prior to and day of dosing (D0-D3)
  * 5mg Olanzapine PO at bedtime or 2.5 mg PO BID on day of dosing (D1, D3)
  Study drug:
  - 60mg Selinexor PO on D1 and D3 of weeks 1-3 of each cycle. Drug holiday on week 4. Courses repeat every 28 days in absence of disease progression or unacceptable toxicity.
Arm/Group | Primary Abiraterone Resistance | Aquired Abiraterone Resistance
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Time to PSA Progression
Description: Time between the first evaluation at which the response criteria are met and the first documentation of PSA (Prostate-Specific Antigen) progression or death. Progression is defined as a rise in PSA of 50% above nadir value or 25% above baseline if there is no decline.
Time Frame: Time between the first evaluation at which the response criteria are met and the first documentation of PSA progression or death or up to 3 years
Measure: Median (Full Range); unit: weeks
Arm/Group | Treatment (Selinexor)
Number analyzed (Participants) | 14
weeks | 12 [7 to 14]

4. Secondary Outcome: Incidence of Non-serious Adverse Events
Description: Incidence of non-serious adverse events, graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0
Time Frame: Up to 3 years after treatment start
Measure: Number; unit: events
Arm/Group | Treatment (Selinexor)
Number analyzed (Participants) | 14
events
  Anorexia | 14
  Hypophosphatemia | 3
  Metabolism and nutrition disorders - Other | 2
  Hypocalcemia | 1
  Hyponatremia | 2
  Weight loss | 7
  Platelet count decreased | 6
  INR increased | 3
  Investigations - Other | 3
  Neutrophil count decreased | 1
  Nausea | 14
  Vomiting | 7
  Constipation | 5
  Diarrhea | 6
  Abdominal distension | 1
  Abdominal pain | 2
  Flatulence | 1
  Gastrointestinal disorders - Other | 1
  Fatigue | 11
  Pain | 3
  Localized edema | 1
  Anemia | 10
  Blood and lymphatic system disorders - Other | 4
  Bone pain | 2
  Pain in extremity | 3
  Arthralgia | 1
  Musculoskeletal/connective tissue disorder, other | 1
  Dizziness | 2
  Presyncope | 3
  Headache | 1
  Hypotension | 5
  Hot flashes | 1
  Blurred vision | 3
  Eye pain | 1
  Night blindness | 1
  Watering eyes | 2
  Lung infection | 1
  Upper respiratory infection | 1
  Urinary tract infection | 1
  Insomnia | 3
  Psychosis | 1
  Cough | 1
  Dyspnea | 1
  Voice alteration | 1
  Cardiac disorders - Other | 1
  Chest pain - cardiac | 1
  Skin and subcutaneous tissue disorders - Other | 2
  Alopecia | 2
  Hematuria | 1

5. Secondary Outcome: Comparison of Leukocyte Exportin 1 (XPO-1) and Macrophage Inhibitory Cytokine-1 (MIC-1) Gene Expression Levels Pre- and Post-Selinexor Treatment
Description: Total RNA isolated from leukocytes of patients will be used for quantitative polymerase chain reaction analysis (qPCR) in order to compare expression levels of XPO-1 and MIC-1 as a function of selinexor dose and total time on treatment.
Time Frame: On days 1 and 15 of course 1 and on day 1 of courses 2 and 3
Population: The study was terminated due to unacceptable toxicity. Data was not collected.
Groups:
- Selinexor Day 1, Course 1; Selinexor Day 15, Course 1; Selinexor Day 1, Course 2; Selinexor Day 1, Course 3: BID: twice a day D: day PO: oral 1 cycle = 4 weeks, 28 days
  Premedication:
  * 8mg Ondansetron PO every 8 hours on day prior to and day of dosing (D0-D3)
  * 5mg Olanzapine PO at bedtime or 2.5 mg PO BID on day of dosing (D1, D3)
  Study drug:
  - 60mg Selinexor PO on D1 and D3 of weeks 1-3 of each cycle. Drug holiday on week 4. Courses repeat every 28 days in absence of disease progression or unacceptable toxicity.
Arm/Group | Selinexor Day 1, Course 1 | Selinexor Day 15, Course 1 | Selinexor Day 1, Course 2 | Selinexor Day 1, Course 3
Number analyzed (Participants) | 0 | 0 | 0 | 0

6. Secondary Outcome: PSA Decline of ≥50% at 12 Weeks Post Therapy Initiation
Description: The number of patients experiencing a PSA decline from baseline of at least 50% in PSA at 12 weeks following the initiation of study therapy.
Time Frame: At 12 weeks post therapy initiation
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Selinexor)
Number analyzed (Participants) | 14
Participants | 1

7. Secondary Outcome: Reduction in Pain for Symptomatic Patients, Measured Using the Brief Pain Inventory (BPI), Short Form
Description: The effect of selinexor on persistent pain associated with bone metastasis, measured using the Brief Pain Inventory (BPI), Short Form. 0 denotes ''no pain'' and 10, ''pain as bad as you can imagine".
Time Frame: At baseline and day 1 of every following cycle until end of treatment or 3 years after study start
Population: The study was terminated due to unacceptable toxicity. Only baseline data was collected.
Measure: Median (Full Range); unit: units on a scale
Groups:
- Pain at Baseline; Pain at Day 1, Course 2 and Following Courses: BID: twice a day D: day PO: oral 1 cycle = 4 weeks, 28 days
  Premedication:
  * 8mg Ondansetron PO every 8 hours on day prior to and day of dosing (D0-D3)
  * 5mg Olanzapine PO at bedtime or 2.5 mg PO BID on day of dosing (D1, D3)
  Study drug:
  - 60mg Selinexor PO on D1 and D3 of weeks 1-3 of each cycle. Drug holiday on week 4. Courses repeat every 28 days in absence of disease progression or unacceptable toxicity.
Arm/Group | Pain at Baseline | Pain at Day 1, Course 2 and Following Courses
Number analyzed (Participants) | 8 | 0
units on a scale | 1.34 [1 to 4] |

8. Secondary Outcome: Serum Selinexor Levels
Description: Serum selinexor trough levels as a function of dose and time since last dose
Time Frame: At day 1 of course 1, each treatment day until end of treatment up to 3 years
Population: The study was terminated due to unacceptable toxicity. Data was not collected.
Arm/Group | Treatment (Selinexor)
Number analyzed (Participants) | 0

9. Secondary Outcome: Time to Confirmed Development of >= 2 New Bone Lesions That Cannot be Attributable to Bone Scan Flare
Description: Defined as time interval between the date of treatment initiation and the date of documented new lesions. Evaluation criteria is defined by the PSAWG2 (Prostate-Specific Antigen Working Group 2) criteria for bone scan evaluation. The time will be 'backdated' to when the >= 2 new lesions were detected if a second scan is done to confirm progression.
Time Frame: At week 8, 16, 24, and every 12 weeks thereafter up to 3 years after treatment start
Population: The study was terminated due to unacceptable toxicity. Data was not collected.
Arm/Group | Treatment (Selinexor)
Number analyzed (Participants) | 0

10. Secondary Outcome: Incidence of Serious Adverse Events
Description: Incidence of serious adverse events, graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0
Time Frame: Up to 3 years after treatment start
Measure: Number; unit: events
Arm/Group | Treatment (Selinexor)
Number analyzed (Participants) | 14
events
  Anemia | 1
  Eye disorders - Other | 2

ADVERSE EVENTS:
Time Frame: 2 years, 6 months
Arm/Group | Treatment (Selinexor)
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 4/14
Other Adverse Events (participants affected / at risk) | 13/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Selinexor) (N=14)
Anemia (Blood and lymphatic system disorders) | 1
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1
Eye disorders - Other, specify (Eye disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Selinexor) (N=14)
Anorexia (Metabolism and nutrition disorders) | 10
Hypophosphatemia (Metabolism and nutrition disorders) | 3
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 2
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Weight loss (Investigations) | 6
Platelet count decreased (Investigations) | 4
INR increased (Investigations) | 1
Investigations - Other, specify (Investigations) | 1
Neutrophil count decreased (Investigations) | 1
Nausea (Gastrointestinal disorders) | 7
Vomiting (Gastrointestinal disorders) | 4
Constipation (Gastrointestinal disorders) | 3
Diarrhea (Gastrointestinal disorders) | 3
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 6
Pain (General disorders) | 2
Localized edema (General disorders) | 1
Anemia (Blood and lymphatic system disorders) | 5
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 2
Presyncope (Nervous system disorders) | 2
Headache (Nervous system disorders) | 1
Hypotension (Vascular disorders) | 5
Hot flashes (Vascular disorders) | 4
Blurred vision (Eye disorders) | 1
Eye pain (Eye disorders) | 2
Night blindness (Eye disorders) | 1
Watering eyes (Eye disorders) | 1
Lung infection (Infections and infestations) | 1
Upper respiratory infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Insomnia (Psychiatric disorders) | 1
Psychosis (Psychiatric disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1
Cardiac disorders - Other, specify (Cardiac disorders) | 1
Chest pain - cardiac (Cardiac disorders) | 1
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 1
Hematuria (Renal and urinary disorders) | 1

LIMITATIONS AND CAVEATS:
The study was terminated due to unacceptable toxicity.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-27): https://cdn.clinicaltrials.gov/large-docs/61/NCT02215161/Prot_SAP_000.pdf